CLINICAL TRIAL: NCT04571944
Title: A Phase 3 Multicenter, Randomized, Placebo-controlled, Double-blind Clinical Study to Evaluate the Efficacy and Safety of MK-4305 (Suvorexant) for Reducing Incidence of Delirium in Japanese Participants at High Risk of Delirium
Brief Title: Efficacy and Safety of Suvorexant (MK-4305) for Reducing Incidence of Delirium in Japanese Participants at High Risk of Delirium (MK-4305-085)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4305-085; MK-4305-085 (Other: MSD); jRCT2031200149 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suvorexant (Experimental): Participants will receive 15 mg of suvorexant orally once daily (QD) for 5 to 7 days.
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): Participants will receive suvorexant-matching placebo orally QD for 5 to 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Suvorexant administered at a dose of 15 mg QD via oral tablet
  Other Names: MK-4305
  Arms: Suvorexant
Drug: Placebo — Suvorexant-matching placebo administered QD via oral tablet
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of suvorexant (MK-4305) for reducing the incidence of delirium in Japanese participants who are at high risk of delirium. The primary hypothesis is that suvorexant reduces the proportion of participants with delirium compared with placebo as assessed by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Is hospitalized for (1) acute disease with severe disease state or decreased daily living function or (2) elective surgery requiring general anesthesia scheduled on the day after or 2 days after admission/Day 1
* Has (1) mild cognitive impairment or mild dementia and/or (2) a history of delirium in any prior hospitalization
* Requires hospitalization for 6 days for acute disease, with treatment starting on day of admission; or 7 days, with treatment starting the day after admission OR
* Requires hospitalization for 6 days for elective surgery scheduled on the day after admission; or for 7 days for elective surgery scheduled 2 days after admission
* Is able to take study medications orally

Exclusion Criteria:

* Has moderate or severe dementia
* Has a history of epilepsy or Parkinson's disease
* Currently uses psychotropic agents or has a mental condition including schizophrenia, other mental disorders, bipolar disorder and major depression
* Has a history of drug or alcohol abuse in the 5 years prior to start of study or has alcoholic disease such as alcoholic liver disease or gastritis alcoholic
* Has a history of narcolepsy or cataplexy
* Has used hypnotics, antipsychotics, mood stabilizers, antidepressants, anxiolytics, psychostimulants, anticonvulsants or tiapride within 2 weeks prior to randomization
* Has delirium as assessed by DSM-5 or DRS-R-98 (total score ≥14.5) before the first dose of study medication

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (50):
- Japan (50):
  - Kohnodai Hospital, National Center for Global Health and Medicine ( Site 8522), Ichikawa, Chiba
  - Iizuka Hospital ( Site 8540), Iizuka, Fukuoka
  - Kokura Memorial Hospital ( Site 8537), Kitakyushu, Fukuoka
  - Maebashi Red Cross Hospital ( Site 8548), Maebashi, Gunma
  - Fukuyama City Hospital ( Site 8528), Fukuyama, Hiroshima
  - Tonan Hospital ( Site 8512), Sapporo, Hokkaido
  - Kansai Rosai Hospital ( Site 8550), Amagasaki, Hyōgo
  - Kanazawa Medical University Hospital ( Site 8514), Kahoku-gun, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center ( Site 8554), Kanazawa, Ishikawa-ken
  - Kagawa University Hospital ( Site 8519), Kita-gun, Kagawa-ken
  - TAKAMATSU Red Cross Hospital ( Site 8547), Takamatsu, Kagawa-ken
  - Nippon Medical School Musashi Kosugi Hospital ( Site 8502), Kawasaki, Kanagawa
  - Showa University Northern Yokohama Hospital ( Site 8534), Yokohama, Kanagawa
  - Yokohama City University Medical Center ( Site 8516), Yokohama, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital ( Site 8541), Yokohama, Kanagawa
  - Yokohama City University Hospital ( Site 8515), Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center ( Site 8531), Yokohama, Kanagawa
  - National Hospital Organization Maizuru Medical Center ( Site 8535), Maizuru-shi, Kyoto
  - Aizawa Hospital ( Site 8542), Matsumoto, Nagano
  - Matsushita Memorial Hospital ( Site 8556), Moriguchi, Osaka
  - Osaka University Hospital ( Site 8524), Suita, Osaka
  - Toyonaka Municipal Hospital ( Site 8521), Toyonaka, Osaka
  - Shimane Prefectural Central Hospital ( Site 8530), Izumo, Shimane
  - Kamitsuga General Hospital ( Site 8546), Kanuma, Tochigi
  - SANO KOSEI GENERAL HOSPITAL ( Site 8551), Sano, Tochigi
  - Jichi Medical University Hospital ( Site 8525), Shimotsuke, Tochigi
  - Yamaguchi University Hospital ( Site 8517), Ube, Yamaguchi
  - National Hospital Organization Kyushu Medical Center ( Site 8532), Fukuoka
  - Gifu Municipal Hospital ( Site 8555), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 8505), Hiroshima
  - National Hospital Organization Kumamoto Medical Center ( Site 8511), Kumamoto
  - Japanese Red Cross Kyoto Daini Hospital ( Site 8533), Kyoto
  - Kyoto Katsura Hospital ( Site 8539), Kyoto
  - Miyazaki Prefectural Miyazaki Hospital ( Site 8543), Miyazaki
  - Niigata City General Hospital ( Site 8544), Niigata
  - Okayama Saiseikai General Hospital ( Site 8549), Okayama
  - Okayama University Hospital ( Site 8510), Okayama
  - Osaka City General Hospital ( Site 8518), Osaka
  - National Hospital Organization Osaka National Hospital ( Site 8536), Osaka
  - Japanese Red Cross Osaka Hospital ( Site 8523), Osaka
  - Nippon Life Hospital ( Site 8552), Osaka
  - Japan Community Health care Organization Osaka Hospital ( Site 8545), Osaka
  - Osaka General Medical Center ( Site 8538), Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 8526), Saga
  - Tokushima Prefectural Central Hospital ( Site 8509), Tokushima
  - National Cancer Center Hospital ( Site 8520), Tokyo
  - National Hospital Organization Tokyo Medical Center ( Site 8529), Tokyo
  - Tokyo Women's Medical University Hospital ( Site 8527), Tokyo
  - Juntendo University Nerima Hospital ( Site 8501), Tokyo
  - Tokyo Medical and Dental University Hospital ( Site 8503), Tokyo

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hatta K, Kishi Y, Wada K, Takeuchi T, Taira T, Uemura K, Ogawa A, Takahashi K, Sato A, Shirakawa M, Herring WJ, Arano I; Suvorexant 085 Study Group. Suvorexant for Reduction of Delirium in Older Adults After Hospitalization: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2427691. doi: 10.1001/jamanetworkopen.2024.27691. PMID 39150711
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant: Participants received 15 mg of suvorexant orally once daily (QD) for 5 to 7 days.
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 105 | 102
Completed | 99 | 102
Not Completed | 6 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — One participant canceled surgery and one participant developed delirium before the first dose. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 105 | 102 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.5 (4.4) | 82.0 (4.9) | 81.7 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 57 | 107
  Male | 55 | 45 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 105 | 102 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 105 | 102 | 207
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Delirium as Assessed by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) Criteria
Description: The DSM-5 is the gold standard for the diagnosis of delirium. DSM-5 criteria were used for clinician assessment of delirium. The percentage of participants with delirium per DSM-5 criteria is presented.
Time Frame: Up to ~8 days
Population: All randomized participants who had at least one assessment of delirium by DSM-5 following administration of at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Groups:
- Suvorexant: Participants received 15 mg of suvorexant orally QD for 5 to 7 days.
- Placebo: Participants received suvorexant-matching placebo orally QD for 5 to 7 days.
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 101 | 102
Percentage of participants | 16.8 | 26.5
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.129, Miettinen and Nurminen method; Analysis was stratified by hospitalization reason (acute disease, elective surgery) and age category (<75 years, ≥75 years); Difference in % vs Placebo = -8.7, 95% CI 2-sided [-20.1 to 2.6]

2. Primary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one or more AEs is presented.
Time Frame: Up to ~21 days
Population: All randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 101 | 102
Participants | 86 | 86
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Other; Difference in % vs. Placebo = 0.8, 95% CI 2-sided [-9.3 to 11.0]

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to ~7 days
Population: All randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 101 | 102
Participants | 2 | 2
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Other; Difference in % vs. Placebo = 0.0, 95% CI 2-sided [-5.1 to 5.2]

4. Secondary Outcome: Maximum Daily Total Score on Delirium Rating Scale-Revised-98 (DRS-R-98)
Description: DRS-R-98 is a diagnostic and assessment tool used for evaluation of delirium. It is a 16-item clinician-rated scale with 13 items measuring delirium severity and 3 diagnostic items. The total DRS-R-98 score can range from 0 (lowest) to 46 (highest). Higher scores indicate worsening or more severe delirium. The maximum daily total score on DRS-R-98 is presented.
Time Frame: Up to ~8 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- Suvorexant: Participants will receive 15 mg of suvorexant orally QD for 5 to 7 days.
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 101 | 102
Score on a scale | 7.0 [4.0 to 13.0] | 7.5 [4.0 to 16.0]
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.485, Hodges-Lehmann method — Based on aligned rank test; Difference vs. Placebo = -0.5, 95% CI 2-sided [-2.0 to 1.0]

5. Secondary Outcome: Percentage of Participants With Delirium as Assessed by DRS-R-98
Description: DRS-R-98 is a diagnostic and assessment tool used for the evaluation of delirium. It is a 16-item clinician-rated scale with 13 items measuring delirium severity and 3 diagnostic items. The total DRS-R-98 score can range from 0 (lowest) to 46 (highest). Higher scores indicate worsening or more severe delirium. Optimized cutoff score for delirium diagnosis in Japanese-translated DRS-R-98 has been determined as ≥14.5. The percentage of participants with delirium as assessed by DRS-R-98, defined as the percentage of participants with total score ≥14.5 per DRS-R-98, is presented.
Time Frame: Up to ~8 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 101 | 102
Percentage of participants | 17.8 | 26.5
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p = 0.136, Miettinen and Nurminen method; [statistical method as in outcome 1, analysis 1]; Difference in % vs. Placebo = -8.6, 95% CI 2-sided [-20.2 to 2.8]

ADVERSE EVENTS:
Time Frame: Up to ~21 days
Description: The safety analysis population included all randomized participants who received at least one dose of study treatment. The analysis population for All-Cause Mortality included all randomized participants.
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 1/105 | 0/102
Serious Adverse Events (participants affected / at risk) | 6/101 | 6/102
Other Adverse Events (participants affected / at risk) | 64/101 | 69/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=101) | Placebo (N=102)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=101) | Placebo (N=102)
Constipation (Gastrointestinal disorders) | 23 (23) | 21 (21)
Nausea (Gastrointestinal disorders) | 8 (8) | 12 (12)
Vomiting (Gastrointestinal disorders) | 13 (13) | 16 (16)
Pyrexia (General disorders) | 4 (4) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 9 (9)
Wound complication (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Delirium (Psychiatric disorders) | 18 (19) | 29 (30)
Insomnia (Psychiatric disorders) | 18 (18) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04571944/Prot_SAP_000.pdf